CLINICAL TRIAL: NCT04882631
Title: A 21 Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of PBI-100 Topical Cream in Healthy Participants Using a Cumulative Irritant Patch Test Design
Brief Title: A Study to Evaluate the Skin Irritation Potential of PBI-100 Topical Cream in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBI-100-101
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: The order of test product patch placement is randomized.
Masking Description: The participant and evaluator are blinded to the identity of the test product (3 strengths of PBI-100), vehicle, negative control and positive control placed on each subject's forearm, upper arm or back
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cumulative Irritation Test (Experimental): Participants will receive topical applications of three concentrations of PBI-100 Topical Cream, one application of vehicle, one application of sodium lauryl sulfate as a positive control and one application of a plain patch as a negative control daily (excluding weekends) for 21 days or 15 applications.
  Interventions: Drug: PBI-100 Topical Cream; Drug: Positive Control - Sodium laurel sulfate (SLS); Other: PBI-100 Topical Cream, Vehicle; Other: Negative Control

INTERVENTIONS:
Drug: PBI-100 Topical Cream — A dose of approximately 560 ug (approximately 0.4 mL of each of the three concentrations to 3 different sites) of PBI-100 was applied daily (excluding weekends) to the skin test sites.
Drug: Positive Control - Sodium laurel sulfate (SLS) — Approximately 0.4 mL of 0.25% SLS was applied daily (excluding weekends) as a positive control test site.
  Other Names: SLS
Other: PBI-100 Topical Cream, Vehicle — Approximately 0.4 mL of 0% placebo cream was applied daily (excluding weekends) as a positive control test site.
Other: Negative Control — A blank patch was applied daily (excluding weekends) as a negative control test site.

SUMMARY:
This is an open-label, single-arm, randomized, evaluator-blinded repeat insult patch testing (RIPT) study wherein test product is applied under an occlusive dressing to the upper back or arm continuously and repeatedly to the same site for a period of 21 days.

DETAILED DESCRIPTION:
This is an open-label, single-arm, randomized, evaluator-blinded repeat insult patch testing (RIPT) study wherein test product is applied under an occlusive dressing to the upper back or arm continuously and repeatedly to the same site for a period of 21 days. Three concentrations of PBI-100 Topical Cream and vehicle (placebo cream) will be applied to the skin of each subject. In addition, one site will be treated with a positive control and another site will be treated with a plain cotton cloth patch and will serve as a negative control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female volunteers between the ages of 18 and 70 years with Fitzpatrick types I, II, or III.
* Must be willing to follow the study requirements and voluntarily give their informed consent.
* Subjects must be able to read and follow study instructions in English.
* Generally in good health as determined by the investigator, based on medical history interview.
* Evidence of a personally signed and dated Informed Consent indicating that the subject has been informed of and understood all pertinent aspects of the trial.

Exclusion Criteria:

* Scars, moles, or other blemishes over the forearm, upper arm, or back that interfere with the study.
* Sunburn within the last three weeks or use of tanning beds.
* History of allergy or hypersensitivity to skin care or consumer products including fragrances, cosmetics, toiletries, or any kind of tape.
* History of chronic or recurrent dermatological diseases, e.g., psoriasis, atopic eczema, chronic urticaria.
* Subjects receiving systemic or topical drugs which can interfere with the development of an inflammatory response, e.g., steroids, immunosuppressive agents, or retinoids.
* History of any significant systemic diseases e.g., cardiac, pulmonary, renal, hepatic, etc. that would impact subject's ability to complete the study.
* Pregnancy or mothers who are breastfeeding or planning a pregnancy.
* Other conditions considered by the Investigator as sound reasons for disqualification from enrollment into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Irritation Potential | 21 days
  Irritation potential based on the Cumulative Irritation Index (CII)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (1):
- KGL Skin Study Center, Newtown Square, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No